CLINICAL TRIAL: NCT01774006
Title: Comparison of Individual Culture and Group Culture of Preimplantation Embryos in Human IVF Treatments
Acronym: GroupCulture
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Peter Fancsovits, Ph.D., Senior Clinical Embryologyst, Semmelweis University
Other Study IDs: SemmelweisU-001
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Other Complications Associated With Artificial Fertilization
Keywords: In vitro fertilization; Embryo transfer; Embryo culture; individual culture; Group culture; embryo quality; Pregnancy rate; Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group culture: Embryos cultured in groups of 2-10
  Interventions: Other: individual embryo culture or group culture
- Individual culture: Embryos cultured individually
  Interventions: Other: individual embryo culture or group culture

INTERVENTIONS:
Other: individual embryo culture or group culture — Embryos cultured in a 25 microliter droplet of culture media individually in a conventional petridish or in groups of 2-10 embryos in a Well-of-the-Well petridish

SUMMARY:
Prospective randomized comparison of two widely used in vitro culture system in human IVF treatments. In vitro fertilized oocytes and embryos are cultured in individual culture media droplets using conventional petridish or in group culture using WOW (well of the well) petridish.

Primary outcome: implantation and pregnancy rates Secondary outcome: fertilization rate and embryo quality

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients entering in vitro fertilization treatment
* at least 1 oocyte collected

Exclusion Criteria:

* no oocytes collected

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients entering in vitro fertilization and embryo transfer treatment
Sampling Method: Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4 weeks after the embryo transfer
  Number of clinical pregnancies (/No. of embryo transfers)
Implantation rate | 4 weeks after embryo transfer
  Number of embryos implanted (/number of embryos transferred)

SECONDARY OUTCOMES:
Fertilization rate | 18 hours after sperm injection
  Number of oocytes fertilized. (only in intracytoplasmic sperm injection cycles)
Embryo quality | 36 and 72 hours after fertilization
  Number and quality of blastomeres, amount of fragmentation embryo grade

OTHER OUTCOMES:
Time needed for evaluation of zygotes and embryos | 18, 24, 36 and 72 hours after fertilization

CONTACTS AND LOCATIONS:
Overall Officials: Janos Urbancsek, DSc, Principal Investigator — Semmelweis University First Department of Obstetrics and Gynecology; Peter Fancsovits, Ph.D., Study Chair — Semmelweis University First Department of Obstetrics and Gynecology; Csaba Pribenszky, Ph.D., Principal Investigator — University of Veterinary Sciences, Budapest; Adam Lehner, MSc, Principal Investigator — Semmelweis University First Department of Obstetrics and Gynecology
Locations (1):
- Semmelweis University First Department of Obstetrics and Gynecology, Budapest, Hungary

REFERENCES:
- [Derived] Fancsovits P, Pribenszky C, Lehner A, Murber A, Kaszas Z, Nemes A, Urbancsek J. Prospective-randomized study comparing clinical outcomes of IVF treatments where embryos were cultured individually or in a microwell group culture dish. Biol Futur. 2022 Jun;73(2):229-236. doi: 10.1007/s42977-022-00113-8. Epub 2022 Mar 12. PMID 35278201